CLINICAL TRIAL: NCT01498770
Title: An Observational Drug Utilization Study of SYCREST^® (Asenapine) in the United Kingdom
Brief Title: An Observational Drug Utilization Study of Asenapine in the United Kingdom (P08308)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P08308; MK-8274-108 (Other: Merck)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine; Aripiprazole; Quetiapine Fumarate; Risperidone; Olanzapine; ziprasidone; iloperidone; Paliperidone Palmitate; Lurasidone Hydrochloride; Clozapine; Amisulpride; sertindole; zotepine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (13):
- Asenapine
  Interventions: Drug: Asenapine
- Aripiprazole
  Interventions: Drug: Aripiprazole
- Quetiapine
  Interventions: Drug: Quetiapine
- Risperidone
  Interventions: Drug: Risperidone
- Olanzapine
  Interventions: Drug: Olanzapine
- Ziprasidone
  Interventions: Drug: Ziprasidone
- Iloperidone
  Interventions: Drug: Iloperidone
- Paliperidone
  Interventions: Drug: Paliperidone
- Lurasidone
  Interventions: Drug: Lurasidone
- Clozapine
  Interventions: Drug: Clozapine
- Amisulpride
  Interventions: Drug: Amisulpride
- Sertindole
  Interventions: Drug: Sertindole
- Zotepine
  Interventions: Drug: Zotepine

INTERVENTIONS:
Drug: Asenapine — Asenapine prescribed as recorded in the CPRD in the UK
  Other Names: Sycrest; SCH 900274
  Groups: Asenapine
Drug: Aripiprazole — Aripiprazole prescribed as recorded in the CPRD in the UK
  Other Names: Abilfy
  Groups: Aripiprazole
Drug: Quetiapine — Quetiapine prescribed as recorded in the CPRD in the UK
  Other Names: Seroquel
  Groups: Quetiapine
Drug: Risperidone — Risperidone prescribed as recorded in the CPRD in the UK
  Other Names: Risperdal
  Groups: Risperidone
Drug: Olanzapine — Olanzapine prescribed as recorded in the CPRD in the UK
  Other Names: Zyprexa
  Groups: Olanzapine
Drug: Ziprasidone — Ziprasidone prescribed as recorded in the CPRD in the UK
  Groups: Ziprasidone
Drug: Iloperidone — Iloperidone prescribed as recorded in the CPRD in the UK
  Groups: Iloperidone
Drug: Paliperidone — Paliperidone prescribed as recorded in the CPRD in the UK
  Groups: Paliperidone
Drug: Lurasidone — Lurasidone prescribed as recorded in the CPRD in the UK
  Groups: Lurasidone
Drug: Clozapine — Clozapine prescribed as recorded in the CPRD in the UK
  Groups: Clozapine
Drug: Amisulpride — Amisulpride prescribed as recorded in the CPRD in the UK
  Groups: Amisulpride
Drug: Sertindole — Sertindole prescribed as recorded in the CPRD in the UK
  Groups: Sertindole
Drug: Zotepine — Zotepine prescribed as recorded in the CPRD in the UK
  Groups: Zotepine

SUMMARY:
This study is designed to describe asenapine prescribing patterns in the United Kingdom (UK) during the post-approval period under conditions of usual practice. The use of asenapine in Bipolar Disorder and other indications will be described. To provide epidemiological and clinical perspective, use of aripiprazole and other comparator drugs will be described.

DETAILED DESCRIPTION:
The data source for this study will be the Clinical Practice Research Database (CPRD) in the UK. New users of asenapine during the period following the UK marketing launch of asenapine will be identified in the CPRD. Use in Bipolar Disorder and other indications, as well as baseline demographic and physical characteristics, including prior health status, comorbidities, concomitant medications and healthcare resource utilization, will be described for the asenapine cohort, for participants aged 18 or greater. Use of asenapine in the general practice setting among pediatric participants will be described.

The primary comparison cohort will be aripiprazole. Participants in the aripiprazole cohort will be matched to participants treated with asenapine based on respective time after market entry. In addition, non-matched cohorts will be used to describe utilization of aripiprazole and other comparators.

ELIGIBILITY:
Inclusion Criteria for Participants Treated with Asenapine:

* At least 1 prescription for asenapine within the study period
* Date of prescription occurs after the CPRD subject registration date or the database specific quality indicator date
* A minimum of 365 or more days of evaluable baseline observation time, occurring prior to the date of prescription for asenapine

Inclusion Criteria for Participants Treated with a Comparator:

* Age 18 years or greater at the time participant receives a prescription for the comparator
* At least 1 prescription for either aripiprazole, quetiapine, risperidone, olanzapine, ziprasidone, iloperidone, paliperidone, lurasidone, clozapine, amisulpride, sertindole or zotepine within the study period
* Date of prescription occurs after the CPRD subject registration date or the database specific quality indicator date
* A minimum of 365 or more days of evaluable baseline observation time, occurring prior to the date of prescription for either aripiprazole, quetiapine, risperidone, olanzapine, ziprasidone, iloperidone, paliperidone, lurasidone, clozapine, amisulpride, sertindole or zotepine

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is drawn from UK general practitioner practices participating in CPRD. The database is generally representative of the UK general population.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Frequency and Proportion of Use, by Psychiatric Diagnosis, Among Asenapine and Aripiprazole Participants Aged 18 or Greater | From baseline through 730 days after date of prescription
Frequency and Proportion of Use Among Asenapine and Aripiprazole Participants Aged 18 or Greater with Schizophrenia and No Diagnosis of Bipolar Disorder | From baseline through 730 days after date of prescription
Frequency and Proportion of Use Among Asenapine and Aripiprazole Participants Aged 18 or Greater with No Diagnosis of Bipolar Disorder or Schizophrenia, by Other Diagnosis | From baseline through 730 days after date of prescription
Baseline Age of Asenapine Participants Aged 18 or Greater Initiating Asenapine During the First Year Since Drug Product Marketing in UK | Baseline observation period (minimum of at least 365 days prior to date of prescription)
Gender of Asenapine Participants Aged 18 or Greater Initiating Asenapine During the First Year Since Drug Product Marketing in UK | Baseline observation period (minimum of at least 365 days prior to date of prescription)
Frequency and Proportion of Pediatric Use, by Psychiatric Diagnosis | From baseline through 365 days after date of prescription
Baseline Age of Asenapine Participants Less Than 18 Years Old Initiating Asenapine During the First Year Since Drug Product Marketing in UK | Baseline observation period (minimum of at least 365 days prior to date of prescription)
Gender of Asenapine Participants Less Than 18 Years Old Initiating Asenapine During the First Year Since Drug Product Marketing in UK | Baseline observation period (minimum of at least 365 days prior to date of prescription)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC